CLINICAL TRIAL: NCT01788475
Title: A Randomized, Pilot Study of the Efficacy and Safety of Ozurdex Steroid Implants in Post-Vitrectomized Eyes in Patients With Diabetic Macular Edema
Brief Title: Safety and Effectiveness of Ozurdex Steroid Implants for DME After Vitrectomy Surgery
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Study withdrawn by Investigator
Sponsor: Lahey Clinic (Other)
Responsible Party: Principal Investigator, Jeffrey L. Marx, MD, Principal Investigator, Lahey Clinic
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2012-031
Record Dates: First submitted 2013-02-07; First posted 2013-02-11 (Estimated); Results first posted 2019-05-08 (Actual); Last update posted 2020-03-12 (Actual); Status verified 2020-03

CONDITIONS: Diabetic Macular Edema
Keywords: Diabetic Macular Edema; DME; Pars Plana Vitrectomy
MeSH Terms: interventions — Dexamethasone; Calcium Dobesilate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Dexamethasone implant up to every 3 Mo. (Active Comparator): Ozurdex (dexamethasone) 0.7 mg implant will be performed on Day 0. All patients will be evaluated monthly thereafter.
  Intervention: One month following initial implantation/sham, patients will be evaluated for focal or grid laser treatment if the investigator feels the patient will benefit.
  Re-implantation of Ozurdex (dexamethasone) may occur at any time > 3 months following last injection in group 1 if any of the following conditions are met:
  1. Increase of > 50 microns from the best previous CRT measurement
  2. Recurrence of intraretinal cystic edema
  3. Persistent intraretinal cystic edema
  Interventions: Drug: Dexamethasone
- Dexamethasone implant up to every 6 Mo. (Active Comparator): Ozurdex (dexamethasone) 0.7 mg implant will be performed on Day 0. All patients will be evaluated monthly thereafter.
  Intervention: One month following initial implantation/sham, patients will be evaluated for focal or grid laser treatment if the investigator feels the patient will benefit.
  Re-implantation of Ozurdex (dexamethasone) may occur at any time >6 months following last injection in group 2 if any of the following conditions are met:
  1. Increase of > 50 microns from the best previous CRT measurement
  2. Recurrence of intraretinal cystic edema
  3. Persistent intraretinal cystic edema
  Interventions: Drug: Dexamethasone
- Sham Implant (Sham Comparator): Sham Procedure will be performed on Day 0. All patients will be evaluated monthly thereafter.
  Intervention: One month following initial implantation/sham, patients will be evaluated for focal or grid laser treatment if the investigator feels the patient will benefit. Also, at 13 months, patients in the sham group will be eligible for Ozurdex (dexamethasone) 0.7 mg implantation if initial inclusion/exclusion criteria are met. These patients would follow re-implantation guidelines of group 2.
  Sham implantation may occur at any time > 6 months following last sham injection in group 3 if any of the following conditions are met:
  1. Increase of > 50 microns from the best previous CRT measurement
  2. Recurrence of intraretinal cystic edema
  3. Persistent intraretinal cystic edema
  Interventions: Drug: Dexamethasone

INTERVENTIONS:
Drug: Dexamethasone — Ozurdex (dexamethasone) 0.7mg steroid implant
  Other Names: Ozurdex; Dexamethasone Posterior segment drug delivery system; DEX PS DDS

SUMMARY:
Currently medications injected intravitreally in previously vitrectomized eyes have a very short half-life due to enhanced clearance of the drug. The use of the Ozurdex (dexamethasone) implant may allow sustained levels of steroid delivery to patients with diabetic macular edema that have undergone prior vitrectomy. The sustained steroid levels may lead to improved central retinal thickness measurements and improved visual acuity.

DETAILED DESCRIPTION:
A total of 15 patients will be enrolled into the study. This is a 3 year randomized controlled study with the primary endpoint at 1 year. Secondary safety and efficacy endpoints will be evaluated in year 2 and year 3.

Patients will be randomly enrolled into 1 of 3 groups:

Group 1: Dexamethasone administered up to every 3 months Group 2: Dexamethasone administered up to every 6 months Group 3: Sham

Patients will be evaluated on a monthly basis with ETDRS visual acuity, intraocular pressure, fundus examination and OCT.

Ozurdex (dexamethasone) or Sham Procedure will be performed on Day 0. All patients will be evaluated monthly thereafter. One month following initial injection/sham, patients will be evaluated for focal or grid laser treatment if the investigator feels the patient will benefit.

Re-implantation of Ozurdex may occur at any time > 3 months following last injection in group 1 and > 6 months following last injection in group 2 if any of the following conditions are met:

1. Increase of > 50 microns from the best previous CRT measurement
2. Recurrence of intraretinal cystic edema
3. Persistent intraretinal cystic edema

At 13 months, patients in the sham group will be eligible for Ozurdex implantation if initial inclusion/exclusion criteria are met. These patients would follow re-implantation guidelines of group 2 (up to every 6 months).

ELIGIBILITY:
Inclusion Criteria:

1. Adults> 18 years of age with type 1 or 2 diabetes mellitus
2. Patients with DME secondary to diabetes mellitus involving the center of the macula OCT thickness is > 300 microns with intraretinal cystic edema
3. BCVA between 20/40 to 20/400
4. Patient had vitrectomy surgery.
5. Provide a signed informed consent prior to any study procedure

Exclusion Criteria:

1. Patient unlikely to benefit from intravitreal Ozurdex due to macular ischemia, atrophy, or other condition
2. Patient with history of steroid response with IOP >35 mm Hg or requirement to be on > 2 glaucoma medications following previous steroid injection.
3. Previous injection of anti-VEGF or steroid in the study eye within 90 days
4. Vitrectomy, cataract surgery, or YAG capsulotomy within 90 days.
5. Current tractional detachment of the macula or vitreous hemorrhage obscuring details of the macula.
6. Pregnant, lactating females, or females of child-bearing potential that are not using reliable contraception.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2013-02-22 (Actual); Primary Completion 2014-11 (Actual); Study Completion 2014-11-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Fina C Barouch, MD, Principal Investigator — Lahey Clinic; Jeffrey L Marx, MD, Study Chair — Lahey Clinic
Locations (1):
- Lahey Medical Center, One Essex Center Drive, Peabody, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Diabetic Retinopathy Clinical Research Network (DRCR.net); Beck RW, Edwards AR, Aiello LP, Bressler NM, Ferris F, Glassman AR, Hartnett E, Ip MS, Kim JE, Kollman C. Three-year follow-up of a randomized trial comparing focal/grid photocoagulation and intravitreal triamcinolone for diabetic macular edema. Arch Ophthalmol. 2009 Mar;127(3):245-51. doi: 10.1001/archophthalmol.2008.610. PMID 19273785
- [Background] Pearson PA, Comstock TL, Ip M, Callanan D, Morse LS, Ashton P, Levy B, Mann ES, Eliott D. Fluocinolone acetonide intravitreal implant for diabetic macular edema: a 3-year multicenter, randomized, controlled clinical trial. Ophthalmology. 2011 Aug;118(8):1580-7. doi: 10.1016/j.ophtha.2011.02.048. PMID 21813090

RESULTS

PARTICIPANT FLOW:
Groups:
- Dexamethasone Implant up to Every 3 Mo.: Ozurdex (dexamethasone) 0.7 mg implant will be performed on Day 0. All patients will be evaluated monthly thereafter.
  Intervention: One month following initial implantation/sham, patients will be evaluated for focal or grid laser treatment if the investigator feels the patient will benefit.
  Re-implantation of Ozurdex (dexamethasone) may occur at any time > 3 months following last injection in group 1 if any of the following conditions are met:
  1. Increase of > 50 microns from the best previous CRT measurement
  2. Recurrence of intraretinal cystic edema
  3. Persistent intraretinal cystic edema
  Dexamethasone: Ozurdex (dexamethasone) 0.7mg steroid implant
- Dexamethasone Implant up to Every 6 Mo.: Ozurdex (dexamethasone) 0.7 mg implant will be performed on Day 0. All patients will be evaluated monthly thereafter.
  Intervention: One month following initial implantation/sham, patients will be evaluated for focal or grid laser treatment if the investigator feels the patient will benefit.
  Re-implantation of Ozurdex (dexamethasone) may occur at any time >6 months following last injection in group 2 if any of the following conditions are met:
  1. Increase of > 50 microns from the best previous CRT measurement
  2. Recurrence of intraretinal cystic edema
  3. Persistent intraretinal cystic edema
  Dexamethasone: Ozurdex (dexamethasone) 0.7mg steroid implant
- Sham Implant: Sham Procedure will be performed on Day 0. All patients will be evaluated monthly thereafter.
  Intervention: One month following initial implantation/sham, patients will be evaluated for focal or grid laser treatment if the investigator feels the patient will benefit. Also, at 13 months, patients in the sham group will be eligible for Ozurdex (dexamethasone) 0.7 mg implantation if initial inclusion/exclusion criteria are met. These patients would follow re-implantation guidelines of group 2.
  Sham implantation may occur at any time > 6 months following last sham injection in group 3 if any of the following conditions are met:
  1. Increase of > 50 microns from the best previous CRT measurement
  2. Recurrence of intraretinal cystic edema
  3. Persistent intraretinal cystic edema
  Dexamethasone: Ozurdex (dexamethasone) 0.7mg steroid implant
Period: Overall Study
Arm/Group | Dexamethasone Implant up to Every 3 Mo. | Dexamethasone Implant up to Every 6 Mo. | Sham Implant
Started | 3 | 0 | 0
Completed | 0 | 0 | 0
Not Completed | 3 | 0 | 0

BASELINE CHARACTERISTICS:
Population: The 3 subjects were withdrawn from the study and returned to standard of care treatment.
Groups:
- Total: Total of all reporting groups
Arm/Group | Dexamethasone Implant up to Every 3 Mo. | Dexamethasone Implant up to Every 6 Mo. | Sham Implant | Total
Number analyzed (Participants) | 3 | 0 | 0 | 3
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 |  |  | 0
  Between 18 and 65 years | 1 |  |  | 1
  >=65 years | 2 |  |  | 2
Age, Continuous [Mean (Standard Deviation); unit: years] | 69 (0) |  |  | 69 (0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 |  |  | 2
  Male | 1 |  |  | 1
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 3 |  |  | 3

OUTCOME MEASURES:

1. Primary Outcome: Visual Acuity Gain
Description: Measured visual acuity gain in number of letters improved as a result of treatment
Time Frame: 13 months
Population: I have entered, "0" into the results section due to the fact that this study was terminated early by the study Principal Investigator and no formal medical record extrapolation, database formation, or analysis was conducted.
Arm/Group | Dexamethasone Implant up to Every 3 Mo. | Dexamethasone Implant up to Every 6 Mo. | Sham Implant
Number analyzed (Participants) | 0 | 0 | 0

2. Secondary Outcome: Central Retinal Thickness Reduction
Description: Central Retinal Thickness Reduction as measured by Heidelberg OCT
Time Frame: 1 year
Population: as for outcome 1
Arm/Group | Dexamethasone Implant up to Every 3 Mo. | Dexamethasone Implant up to Every 6 Mo. | Sham Implant
Number analyzed (Participants) | 0 | 0 | 0

3. Secondary Outcome: Comparison of Efficacy Between Group 1 and 2
Description: Comparison of efficacy between group 1 and group 2
Time Frame: 3 years
Population: as for outcome 1
Arm/Group | Dexamethasone Implant up to Every 3 Mo. | Dexamethasone Implant up to Every 6 Mo. | Sham Implant
Number analyzed (Participants) | 0 | 0 | 0

4. Secondary Outcome: Visual Acuity Gain at Year 2 and 3
Description: VA gain in ETDRS letters at years 2 and years 3
Time Frame: 3 years
Population: as for outcome 1
Arm/Group | Dexamethasone Implant up to Every 3 Mo. | Dexamethasone Implant up to Every 6 Mo. | Sham Implant
Number analyzed (Participants) | 0 | 0 | 0

5. Secondary Outcome: Time to Reimplantation of Ozurdex Implant
Description: Time in months until new implant is needed
Time Frame: 3 years
Population: as for outcome 1
Arm/Group | Dexamethasone Implant up to Every 3 Mo. | Dexamethasone Implant up to Every 6 Mo. | Sham Implant
Number analyzed (Participants) | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: Baseline through study termination.
Description: This study was terminated early by the study Principal Investigator. All 3 subjects were enrolled in the study, but were converted to standard of care less than 6 months from enrollment.
Arm/Group | Dexamethasone Implant up to Every 3 Mo. | Dexamethasone Implant up to Every 6 Mo. | Sham Implant
All-Cause Mortality (participants affected / at risk) | 0/3 | 0/0 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/3 | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/3 | 0/0 | 0/0

LIMITATIONS AND CAVEATS:
The study was terminated early leading to small numbers of subjects analyzed.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days